CLINICAL TRIAL: NCT06696300
Title: Comparison of the Effects of Foundation and Functional Inspiratory Muscle Training in Addition to Classical Physiotherapy in Non-Specific Chronic Low Back Pain
Brief Title: Effects of Foundation and Functional Inspiratory Muscle Training in Non-Specific Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Collaborators: Hacettepe University (Other); Selcuk University (Other)
Responsible Party: Principal Investigator, Fatih ÖZYURT, Physiotherapist, Research Assistant, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/19
Record Dates: First submitted 2024-11-13; First posted 2024-11-20 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain, Mechanical; Low Back Pain, Chronic; Non Specific Chronic Low Back Pain
Keywords: Low Back Pain; Respiratory Muscle Strength; Muscle Training; Classical Physiotherapy; Ultrasound
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluations will be made by a single evaluator who is unaware of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classical Physiotherapy Group (Active Comparator)
  Interventions: Other: Classical Physiotherapy Group
- Foundation Inspiratory Muscle Training (Experimental)
  Interventions: Other: Classical Physiotherapy Group; Other: Foundation Inspiratory Muscle Training in Addition to Classical Physiotherapy
- Functional Inspiratory Muscle Training Group (Experimental)
  Interventions: Other: Classical Physiotherapy Group; Other: Functional Inspiratory Muscle Training Group in Addition to Classical Physiotherapy

INTERVENTIONS:
Other: Classical Physiotherapy Group — Classical physiotherapy group (CF) will be treated face to face for 30 sessions in total, 3 days a week, 10 weeks. Hotpack, Ultrasound, TENS and Basic Exercises will be applied to the CF group. Hotpack will be applied superficially to the lumbar region for 15 minutes. Ultrasound 1MHz- 1.5 Wt/cm2 will be applied to the lumbar region. TENS 50 Hz will be applied for 15 minutes, leaving the painful area in the middle. Basic exercises will be applied as 8-12 repetitions, 2 sets. The number of repetitions and sets will be increased as the tolerance of the patients increases.
  Pelvic tilt exercises Supine hip flexor stretch Supine lumbar extensor stretch Crunches Cat-Camel Exercises
Other: Foundation Inspiratory Muscle Training in Addition to Classical Physiotherapy — In addition to Classical Physiotherapy, Foundation Inspiratory Muscle Training (IKE) will be treated face to face for 30 sessions, 3 days a week, 10 weeks. On other days, IKE will be applied at home for 15 minutes in the morning and evening for a total of 30 minutes and will be followed up with a diary. IKE will be applied with a device that can load with threshold pressure. The IKE group will continue the exercise program for 10 weeks. The intensity of the exercise will be adjusted to 40-50% MIP for the exercise group. After 10 consecutive respiratory cycles, 3-4 respiratory controls will be asked. As tolerance increases, the consecutive respiratory cycle will be increased. The intensity will be adjusted by taking weekly MIP measurements. Daily monitoring forms will be created for each participant to ensure exercise follow-up.
  Arms: Foundation Inspiratory Muscle Training
Other: Functional Inspiratory Muscle Training Group in Addition to Classical Physiotherapy — Functional Inspiratory Muscle Training Group will receive functional inspiratory muscle training in addition to classical physiotherapy, 3 days a week, 10 weeks, 30 sessions in total, face-to-face treatment. On other days, foundation-ICE will be applied at home for 15 minutes in the morning and evening, for a total of 30 minutes, and will be followed with a diary. The same protocol will be applied with the foundation IKE group for teaching the respiratory cycle in the first 4 weeks, and resisted breathing will be worked simultaneously with the exercises in Table 2 in the last 6 weeks. The exercise program will be continued for a total of 10 weeks, including F-ICE, foundation IKE for the first 4 weeks, and F-ICE for 6 weeks thereafter. The intensity of the exercise will be adjusted to 40-50% MIP for the exercise group. After 10 consecutive respiratory cycles, 3-4 respiratory controls will be requested. As tolerance increases, the number of consecutive respiratory cycles will be increase
  Arms: Functional Inspiratory Muscle Training Group

SUMMARY:
This study was planned to examine the effects of basic and functional respiratory muscle training on pain, disability level, and functionality. In this study, participants will be randomly divided into 3 groups. The first group will be treated with physical therapy applications applied in state hospitals for 10 weeks. The second group will receive basic respiratory muscle training treatment in addition to physical therapy in state hospitals. The third group will receive respiratory muscle training with exercise in addition to physical therapy in state hospitals. Evaluations will be made before the first session, after the 30th session, in the 3rd month, in the 6th month, and in the 1st year. There is no interventional method in the evaluations. Pain intensity, disability level, physical activity status, quality of life, fear of movement, pain catastrophizing, anxiety and depression levels will be questioned with scales. In physical measurements, participant's aerobic capacity will be measured with the 2-Minute Walk Test, participants's flexibility with the sit-and-long test, participants's respiratory muscle strength with the MIP/MEP device, participants's core endurance with the trunk flexor muscle endurance test, participants's lower and upper extremity muscle strength with a handheld dynamometer, participants's postural control with the Biodex balance device, and participants's muscle thickness with an ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being between the ages of 18-65,
* Having low back pain that has been ongoing for at least 3 months (12 weeks),
* Having a Visual Analog Scale (VAS) of pain intensity of ≥3,
* Being right-hand dominant.

Exclusion Criteria:

* Not volunteering to participate in the study,
* Having a history of cancer,
* Having a spinal infection,
* Having a rheumatological condition,
* Having a spinal fracture,
* Having red flag signs (sudden and unexpected weight loss, fever, etc.)
* Having a psychological disorder,
* Having a previous spinal surgery,
* Having radiculopathy (neuropathic pain along the lower extremity due to nerve root compression),
* Not continuing home exercises more than 80%,
* Having an anatomical and congenital abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Sociodemographic Information | Baseline
  Participants' sociodemographic information form will include body weight (kilogram).
Evaluation of Sociodemographic Information | Baseline
  Participants' sociodemographic information form will include, height (centimeter).
Evaluation of Sociodemographic Information | Baseline
  Participants' sociodemographic information form will include gender (male/female), age (years), dominant upper extremity (hand with which to eat), location of pain (middle, right, left), severity of pain (VAS), level of education, profession, occupational activity status, exercise habits (yes/no), alcohol and cigarette consumption (yes/no), family history, personal history, accompanying illnesses and medications used. Participants' body mass indexes will be calculated using the kg/m2 formula and recorded.
Assessment of Pain Intensity | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  Pain intensity will be measured with Visual Analog Scale (VAS). VAS asks the patient to mark the intensity of pain he/she has felt during the past week between 0-10 cm (0- I have no pain, 10- I have the most severe pain I can feel). High scores indicate severe pain. VAS is a valid and reliable method for determining the intensity of pain in individuals with NSCLBP.
Evaluation of Disability Level | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  The level of disability will be assessed with the Oswetry Disability Index (ODI). The level of disability due to back pain in patients with limitations in their daily lives and functional movements was assessed with the ODI. The ODI, consisting of 10 questions, questions the patients' travel activities, sexual life, sleep, social life, sitting, walking, standing, pain intensity, lifting and personal care activities. Each question is scored between 0-5 (0- Does not interfere at all, 5- Completely interferes). High scores indicate a high level of disability.
Respiratory Muscle Strength Assessment | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  Respiratory muscle strength will be measured before and after interventions for peripheral muscle strength. Respiratory muscle strength will be measured with a portable device (Intraoral pressure measuring device) that can measure intraoral pressure electronically. Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be recorded with intraoral pressure measurement, which is a non-invasive method .
Diaphragm, Transversus abdominis and Multifidus, Muscle Thickness Evaluation | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  Diaphragm thickness and mobility will be evaluated with ultrasonography Clarius C3HD, (Clarius Mobile Health, BC, Canada). Diaphragm thickness measurements will be made using 8-15 mHz linear probe from 8-9th intercostal space. Functional residual capacity (FRC) level will be measured at the end of maximum expiration and total lung capacity (TLC) level will be measured at the end of maximum inspiration. Thickening ratio will be calculated using end-inspiratory diaphragm thickness/end-expiratory diaphragm thickness formula, and thickening fraction will be calculated using end-inspiratory thickness-end-expiratory thickness/end-expiratory thickness formula. Diaphragm mobility will be evaluated using M-mode during rest and deep inspiration with 1-6 mHz convex probe.

SECONDARY OUTCOMES:
Physical Activity Assessment | Baseline
  Physical activity will be assessed using the short form of the International Physical Activity Questionnaire (SFIPAQ). The seven-question questionnaire lists activities and asks about the duration and frequency of each activity during the past week. The MET values defined for walking (3.3 METs), moderate-intensity physical activity (4.0 METs), and vigorous-intensity physical activity (8.0 METs) are multiplied by the duration (minutes) and frequency (days) to calculate the physical activity score in terms of "MET-min/week". The question of sitting is not included in the physical activity score (103). Physical activity levels will be classified as inactive (<600 MET-min/week), minimally active (600-3000 MET-min/week), and active (>3000 MET-min/week).
Evaluation of Exercise Capacity | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  Exercise capacity will be assessed with the "2-Minute Walk Test (2MWT)" before and after the interventions. The 2MWT is a frequently used, low-cost, clinically significant and recommended test for the assessment of functional exercise capacity. During the test, the person is asked to walk as fast as possible for two minutes in a 15-meter corridor. Before the test, the person is informed that they can stop and rest whenever they want, but this time will not be added. During the test, the person will be encouraged using standard expressions every minute. After the test, the total distance walked is recorded in meters.
Evaluation of Flexibility | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  The patient's flexibility will be assessed with the sit and reach test. The patient will be positioned with one foot resting on the S&R Sit and Reach® measuring table, the sole of the other foot on the floor, and the leg bent at the knee. The patient performing the application will place their hands on top of each other and stretch forward slowly and in a controlled manner. Then, the therapist will ask them to reach out with their hands on the S&R Sit and Reach® ruler three times and record the best degree. The data will be recorded in centimeters .
Lower and Upper Extremity Muscle Strength | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  Patients' knee extensor and shoulder abductor muscle strengths will be measured using a portable handheld dynamometer. Measurements will be repeated three times for the dominant and non-dominant sides, and the highest values will be recorded in kgF.
Core Endurance Assessment | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  The trunk flexor endurance test will be used to assess core endurance. Before the test begins, the head of the bed will be brought to 60°. The participant will lean their back against the head of the bed and then bring their knees and hips to 90° flexion. During this time, the participant's upper extremities will be crossed on the chest. With the start of the test, the head of the bed will be lowered and the participant will be asked to maintain their position. The time the participant spends without changing their position will be noted in seconds. The test will be repeated once.
Postural Control Evaluation | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  Postural control will be evaluated with the Biodex® system, which is actively used in our clinic before and after the interventions. Increasing scores in the Biodex Balance System indicate that balance is deteriorating. After a 20-second trial period for statics, they will be asked to keep the circular ring in the center by moving it in the anteroposterior and mediolateral directions. Level 6 of the 8-level resistance (1 is the least stable, 8 is the most stable) will be used in the evaluation of dynamic balance. At the end of the 20-second test period, the general stability index, anteroposterior stability index, mediolateral stability index and general stability index scores of all individuals will be recorded for both static and dynamic balance.
Evaluation of Quality of Life | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  Short Form-12 consists of 8 sub-dimensions and 12 items: physical functioning (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functioning (1 item), emotional role (2 items) and mental health (2 items). While the items related to physical and emotional role are answered as dichotomous (yes or no), other items have Likert-type options ranging from 3 to 6. The total score of the survey varies between 0-100, with higher scores representing better health.
Fear of Movement | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  The Tampa Kinesiophobia Scale (TKS) is a 17-question checklist used to assess acute and chronic low back pain, fibromyalgia, and musculoskeletal injuries and whiplash-related conditions. The scale uses a 4-point Likert scale (1 = Strongly disagree, 4 = Strongly agree). A total score is calculated after items 4, 8, 12, and 16 are reversed. The individual receives a total score between 17 and 68. A high score on the scale indicates that the individual has high kinesiophobia.
Pain Catastrophizing | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  Pain catastrophizing of patients will be assessed using the "Pain Catastrophizing Scale (PCS)". The Turkish version of the "Pain Catastrophizing Scale", which has been reported to reliably predict certain variables such as fear, emotion or thought related to individuals' past pain experiences, severe pain, disability and emotional disturbances, will be assessed using the Pain Catastrophizing Scale (PCS). The scale consists of 13 questions scored from 0 to 4 (0=Not at all, 1=Somewhat. 2=Moderately, 3=Severely, 4=Always). An increase in the scale score indicates a high fear of experiencing pain .
Anxiety and Depression | Baseline- 10 weeks- 3 Months- 6 Months- 1 Year
  The Hospital Anxiety and Depression Scale is used to determine the risk of anxiety and depression in patients and to measure their levels and changes in severity. The scale consists of a total of 14 questions. Seven of these (odd numbers) measure anxiety, and the other seven (even numbers) measure depression. The scale provides a four-point Likert-type measurement. Each item is scored differently. Items 1, 3, 5, 6, 8, 10, 11 and 13 are in decreasing severity and are scored as 3, 2, 1, 0. Items 2, 4, 7, 9, 12 and 14 are scored as 0, 1, 2, 3. The total scores of the subscales are obtained by adding these item scores. While items 1, 3, 5, 7, 9, 11 and 13 are added for the anxiety subscale, the scores of items 2, 4, 6, 8, 10, 12 and 14 are added for the depression subscale. Each heading is scored from 0 to 21. Higher scores indicate higher anxiety and depression.
Treatment Satisfaction | 10 weeks
  Treatment satisfaction will be assessed with VAS. The patient will be asked to mark their level of satisfaction after treatment between 0-10 cm. A high score will indicate a high level of satisfaction.
Willingness for Treatment | Baseline
  Willingness for treatment will be assessed with VAS. The patient will be asked to mark their willingness level between 0-10 cm before treatment. A high score will indicate a high level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Akbayrak, Professor, Study Director — Hacettepe University
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kolar P, Sulc J, Kyncl M, Sanda J, Cakrt O, Andel R, Kumagai K, Kobesova A. Postural function of the diaphragm in persons with and without chronic low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):352-62. doi: 10.2519/jospt.2012.3830. Epub 2011 Dec 21. PMID 22236541
- [Result] Janssens L, Brumagne S, Polspoel K, Troosters T, McConnell A. The effect of inspiratory muscles fatigue on postural control in people with and without recurrent low back pain. Spine (Phila Pa 1976). 2010 May 1;35(10):1088-94. doi: 10.1097/BRS.0b013e3181bee5c3. PMID 20393397
- [Result] Finta R, Nagy E, Bender T. The effect of diaphragm training on lumbar stabilizer muscles: a new concept for improving segmental stability in the case of low back pain. J Pain Res. 2018 Nov 28;11:3031-3045. doi: 10.2147/JPR.S181610. eCollection 2018. PMID 30568484
- [Result] Calvo-Lobo C, Almazan-Polo J, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Palomo-Lopez P, Rodriguez-Sanz D, Lopez-Lopez D. Ultrasonography comparison of diaphragm thickness and excursion between athletes with and without lumbopelvic pain. Phys Ther Sport. 2019 May;37:128-137. doi: 10.1016/j.ptsp.2019.03.015. Epub 2019 Mar 28. PMID 30954705